CLINICAL TRIAL: NCT01922362
Title: The Use of "Negative Pressure Drainage System" for Caring Split-thickness Skin Graft Recipient Sites
Brief Title: Negative Pressure Drainage System Split-thickness Skin Graft Recipient Sites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-12-022B
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Wound Healing of STSG
Keywords: STSG; wound healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Negative pressure drainage system (Experimental): Negative pressure drainage system
  Interventions: Device: Negative pressure drainage system
- Indirect wet dressing group (Active Comparator): Indirect wet dressing
  Interventions: Device: Indirect wet dressing

INTERVENTIONS:
Device: Negative pressure drainage system — a close system surgical drain was placed over the graft with the length equal to the wound size. A silicon penrose drain with side holes on it covered the surgical drain to prevent direct contact of transparent film and the surgical drain, which led to poor drainage function. The penrose drains were excluded from the system during the test period due to the same function of a close system surgical drain with and without a penrose drain. A transparent film was place over the graft and drains and over a margin of the surrounding healthy skin.
  Arms: Negative pressure drainage system
Device: Indirect wet dressing — The recipient site wound is covered with sulfa-tula first and then wet gauze.
  Arms: Indirect wet dressing group

SUMMARY:
To compare the efficacy and safety of negative pressure drainage system with controls (indirect saline soaks) in the coverage of recipient site wounds of split-thickness skin graft.

DETAILED DESCRIPTION:
Randomized, comparator-controlled trial in patients underwent split-thickness skin graft conducted in Taipei Veterans General Hospital between Aug. 2012 and Dec. 2013. (No.) patients age 21 to 60 years were randomly assigned in the intervention group (n= ) of negative pressure drainage system or to a control group (n= ) of traditional method. Patients who had immunologic disease, end-stage renal disease, coagulopathy, or history of radiation were excluded. The conditions of graft take and pain and discomfort were compared every day during the first 7 days after operation and 2 weeks and 3 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 60 years
* The wounds located on limbs or trunk
* The area of wounds is ranged 50 to 250cm2.

Exclusion Criteria:

* immunodeficiency disease
* end stage renal disease
* coagulopathy
* history of radiation to the recipient site
* allergy to the dressing
* major medical problems

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Healing of the wound at the 7th day after operation | 1 week

SECONDARY OUTCOMES:
Pain, Comfort, and satisfication of the device | one week
Long term wound condition | three months
  Such as area of non-healing, erosion, infection, or scar hypertrophy

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veteran General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] WINTER GD. Formation of the scab and the rate of epithelization of superficial wounds in the skin of the young domestic pig. Nature. 1962 Jan 20;193:293-4. doi: 10.1038/193293a0. No abstract available. PMID 14007593
- [Background] HINMAN CD, MAIBACH H. EFFECT OF AIR EXPOSURE AND OCCLUSION ON EXPERIMENTAL HUMAN SKIN WOUNDS. Nature. 1963 Oct 26;200:377-8. doi: 10.1038/200377a0. No abstract available. PMID 14087904
- [Background] Vogt PM, Andree C, Breuing K, Liu PY, Slama J, Helo G, Eriksson E. Dry, moist, and wet skin wound repair. Ann Plast Surg. 1995 May;34(5):493-9; discussion 499-500. doi: 10.1097/00000637-199505000-00007. PMID 7639486
- [Background] Christian MM, Behroozan DS, Moy RL. Delayed infections following full-face CO2 laser resurfacing and occlusive dressing use. Dermatol Surg. 2000 Jan;26(1):32-6. doi: 10.1046/j.1524-4725.2000.99042.x. PMID 10632683
- [Background] Wang TH, Ma H, Yeh FL, Lin JT, Shen BH. The use of "composite dressing" for covering split-thickness skin graft donor sites. Burns. 2010 Mar;36(2):252-5. doi: 10.1016/j.burns.2009.04.003. Epub 2009 Jun 7. PMID 19505763
- [Background] Alvarez OM, Mertz PM, Eaglstein WH. The effect of occlusive dressings on collagen synthesis and re-epithelialization in superficial wounds. J Surg Res. 1983 Aug;35(2):142-8. doi: 10.1016/0022-4804(83)90136-1. PMID 6887836
- [Background] Nemeth AJ, Eaglstein WH, Taylor JR, Peerson LJ, Falanga V. Faster healing and less pain in skin biopsy sites treated with an occlusive dressing. Arch Dermatol. 1991 Nov;127(11):1679-83. PMID 1952972
- [Background] Scherer SS, Pietramaggiori G, Mathews JC, Prsa MJ, Huang S, Orgill DP. The mechanism of action of the vacuum-assisted closure device. Plast Reconstr Surg. 2008 Sep;122(3):786-797. doi: 10.1097/PRS.0b013e31818237ac. PMID 18766042
- [Background] Petkar KS, Dhanraj P, Kingsly PM, Sreekar H, Lakshmanarao A, Lamba S, Shetty R, Zachariah JR. A prospective randomized controlled trial comparing negative pressure dressing and conventional dressing methods on split-thickness skin grafts in burned patients. Burns. 2011 Sep;37(6):925-9. doi: 10.1016/j.burns.2011.05.013. Epub 2011 Jul 1. PMID 21723044
- [Background] Li TS, Choong MY, Wu HF, Chung KC. Simplified negative-pressure wound therapy system for skin graft wounds. Plast Reconstr Surg. 2012 Feb;129(2):399e-401e. doi: 10.1097/PRS.0b013e31823af1a8. No abstract available. PMID 22286487